CLINICAL TRIAL: NCT02788838
Title: The Impact of Food Advertisements on Brain Response and Eating Behavior in Children
Status: Completed | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kathleen Loralee Keller, Assistant Professor, Penn State University
Other Study IDs: CommercialEating01
Record Dates: First submitted 2016-05-24; First posted 2016-06-02 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Pediatric Obesity
Keywords: Magnetic Resonance Imaging; Energy Intake; Commercials; Children
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this project is to examine the impact that television food advertisements have on brain responses and eating behavior in children. Food advertisements enhance children's liking and intake of foods that tend to be high in energy content and low in nutritional value. Although several studies have measured the differences in children's food intake after watching advertisements, none have shown the brain mechanisms associated with this change in behavior. In order to clarify the relationship between food advertising and eating behavior, the investigators have assembled a team with expertise in functional imaging, eating behaviors, and clinical pediatric research. First, the investigators will observe the differences in children's eating behaviors after being exposed to food commercials or non-food commercials. Second, the investigators will measure the difference in child brain response to high and low energy foods after being exposed to food commercials or non-food commercials. These data will allow us to identify which areas of the brain are specifically affected by exposure to food commercials and correlate activity in these areas with children's measured food intake in the laboratory. Children ages 7-9 will participate in this 5-visit study which will be completed over the course of 12 months. Understanding how food advertisements impact children's brain responses and subsequent eating behaviors will have implications for understanding why some children respond differently to these cues than others. These outcomes may also inform the development of more effective programs and policies to prevent childhood obesity.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* English as native language
* Reading at/above grade level
* Not Claustrophobic
* Generally Healthy

Exclusion Criteria:

* Left-handedness
* Metal in or on body that cannot be removed
* Claustrophobic
* Medication usage that may alter brain activity or blood flow
* Medical disorder that may impact comfort or safety in MRI scanner
* Food allergies

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children ages 7-9 years old
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI), blood oxygen level dependent (BOLD) response to high and low energy foods following food commercial priming | Collected at fMRI scan at week 4 or 5 (randomized)
  Whole-brain response to food images varied by 2 levels of energy viewed in 2 conditions
Functional magnetic resonance imaging, blood oxygen level dependent (BOLD) response to high and low energy foods following toy commercial priming | Collected at fMRI scan at week 4 or 5 (randomized)
  Energy intake of foods consumed ad libitum at each laboratory test-meal in 3 conditions
Baseline Energy Intake | Collected at week 1 of the study
  Energy intake of foods consumed ad libitum at laboratory test-meal with no priming stimulus
Energy Intake following food commercials | Collected at week 2 or 3 (randomized) of the study
  Energy intake of foods consumed ad libitum at laboratory test-meal following food commercials priming
Energy Intake following toy commercials | Collected at week 2 or 3 (randomized) of the study
  Energy intake of foods consumed ad libitum at laboratory test-meal following toy priming stimulus

SECONDARY OUTCOMES:
Region of Interest (ROI)-response to food type by condition | Collected at fMRI scans at weeks 4 and 5 of study
  Response in selected regions of interest to images varied by 2 levels of energy viewed in 2 conditions

OTHER OUTCOMES:
Appetitive traits | Collected at week 1
  Parent-reported questionnaire of habitual eating styles in children
Television and Internet use and exposure | Collected at week 1
  Parent and child reported questionnaires of television and internet use and exposure to shows and commercials
BMI-z score | Collected at week 1
  BMI-z score calculated using age, sex, weight, and height
Liking and Wanting of Foods | Collected at week 1
  Ratings to how much child likes and wants specific foods used in the test meals on child friendly computerized rating scale
Pubertal Development | Collected at week 1
  Parent reported pubertal development through questionnaire
Parental feeding strategies | Collected at week 1
  Parent-reported measures of feeding practices
Height | Collected at week 1
  Height in cm measured by stadiometer
Weight | Collected at week 1
  Weight in kg measured by standard digital scale
Body Fat Percentage | Collected at week 1
  Body Fat Percentage assessed by Bio Electrical Impedance Scale
BMI | Collected at week 1
  Calculated from height and weight (kg/m^2)

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States